CLINICAL TRIAL: NCT00742885
Title: Immunogenicity and Safety of GSK Biologicals' (Pre-) Pandemic Influenza Candidate Vaccine GSK 1557484A.
Brief Title: Immunogenicity and Safety of GSK Biologicals' (Pre-) Pandemic Influenza Candidate Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 111756
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Immunogenicity; Safety; Pandemic Influenza
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Influenza A (H5N1) 20-40 Years Group (Experimental): Subjects aged between 20 and 40 years inclusive received 2 doses of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted at Days 0 and 21 administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted
- Influenza A (H5N1) 41-64 Years Group (Experimental): Subjects aged between 41 and 64 years inclusive received 2 doses of Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted at Days 0 and 21 administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted

INTERVENTIONS:
Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted — All subjects will receive 2 doses administered as an intramuscular (IM) injection.
  Other Names: PumarixTM

SUMMARY:
This trial will assess the immunogenicity and safety elicited by the adjuvanted GSK Biologicals' (pre-) pandemic influenza candidate vaccine in healthy Japanese adults.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male and female adults 20 to 64 years of age at time of the first vaccination, inclusive.
* Good general health as assessed by medical history and physical examination.
* Access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device.
* Written informed consent obtained from the subject.
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.

Exclusion Criteria:

* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness.
* Presence or evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Diagnosed with cancer, or treatment for cancer within 3 years.
* Presence of an axillary temperature >= 37.5 °C, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Receipt of systemic glucocorticoids within 1 month of study enrolment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrolment.
* Any significant disorder of coagulation or treatment with Coumadin derivatives or heparin.
* Administration of any registered vaccine within 30 days before study enrolment or planned administration within the first vaccination up to blood sampling at Day 42 and within 30 days prior to blood sampling at Day 182.
* Use of any investigational or non-registered product within 30 days prior to study enrolment or planned use during the study period.
* History of previous H5N1 vaccination, or history of H5N1 influenza infection.
* Receipt of any immunoglobulins and/or any blood products within 6 months of study enrolment or planned administration of any of these products during the study period.
* Any known or suspected allergy to any constituent of influenza vaccines or component used in the manufacturing process of the study vaccine, a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin test result prior to the time of first vaccination.
* Lactating or nursing.
* Women of child-bearing potential who lack a history of reliable contraceptive practices. The provision of this history does NOT replace the requirement to perform, and obtain negative results in pregnancy urine tests prior to treatments; all women will have urine pregnancy tests regardless of their status.
* Known receipt of analgesic or antipyretic medication on the day of treatment (Day 0).

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2008-09-01; Primary Completion 2009-03-07 (Actual); Study Completion 2009-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Japan (2):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Nagai H, Ikematsu H, Tenjinbaru K, Maeda A, Drame M, Roman FP. A phase II, open-label, multicentre study to evaluate the immunogenicity and safety of an adjuvanted prepandemic (H5N1) influenza vaccine in healthy Japanese adults. BMC Infect Dis. 2010 Nov 25;10:338. doi: 10.1186/1471-2334-10-338. PMID 21108818
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111756 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Started | 50 | 50
Completed | 49 (to Day 182) | 50 (to Day 182)
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.1 (5.69) | 49.6 (6.04) | 40.3 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 32 | 57
  Male | 25 | 18 | 43

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers for the H5N1 Vaccine Strain
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The H5N1 vaccine strain included A/Indonesia/05/2005 antigen (A/Indonesia).
Time Frame: At Day 0 and Day 42
Population: Analysis was performed on According-To-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and assay results were available for antibodies against the study vaccine antigen component after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Titer
  A/Indonesia at Day 0 | 5.0 [5.0 to 5.0] | 5.4 [5.0 to 5.8]
  A/Indonesia at Day 42 | 156.8 [105.8 to 232.3] | 142.1 [104.0 to 194.3]

2. Primary Outcome: Number of Subjects Seroconverted for H5N1 HI Antibodies
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer. The H5N1 vaccine strain included A/Indonesia antigen.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants | 45 | 46

3. Primary Outcome: HI Antibody Seroconversion Factors for H5N1 HI Antibodies
Description: Seroconversion factors (SCF) were defined as the fold increase in serum H5N1 HI antibody GMTs post-vaccination compared to Day 0, at Day 42. The H5N1 vaccine strain included A/Indonesia antigen.
Time Frame: At Day 0 and Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Fold Increase | 31.4 [21.2 to 46.5] | 26.2 [19.2 to 35.8]

4. Primary Outcome: Number of Subjects Seroprotected for H5N1 HI Antibodies
Description: A seroprotected subject was defined as a subject with a serum H5N1 HI antibody titer greater than or equal to 1:40, at Day 42. The H5N1 vaccine strain included A/Indonesia antigen.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants | 45 | 46

5. Primary Outcome: Haemagglutination Inhibition (HI) Antibody Titers for the H5N1 Vaccine Strain
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The H5N1 vaccine strain included A/Indonesia antigen.
Time Frame: At Day 0, Day 21 and Day 182
Population: Analysis was performed on According-To-Protocol (ATP) cohort for persistence which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and assay results were available for antibodies against the study vaccine antigen component on Day 182.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Titer
  A/Indonesia at Day 0 | 5.0 [5.0 to 5.0] | 5.4 [5.0 to 5.8]
  A/Indonesia at Day 21 | 15.8 [11.0 to 22.8] | 15.4 [10.7 to 22.0]
  A/Indonesia at Day 182: number analyzed (Participants) | 49 | 50
  A/Indonesia at Day 182 | 25.6 [17.3 to 38.1] | 37.4 [27.5 to 50.8]

6. Secondary Outcome: Number of Subjects Seroconverted for H5N1 HI Antibodies
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a pre-vaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer, at Days 21 and 182. The H5N1 vaccine strain included A/Indonesia antigen.
Time Frame: At Day 21 and Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  A/Indonesia at Day 21 | 19 | 16
  A/Indonesia at Day 182: number analyzed (Participants) | 49 | 50
  A/Indonesia at Day 182 | 29 | 38

7. Secondary Outcome: Seroconversion Factors for H5N1 HI Antibodies
Description: Seroconversion factors (SCF) were defined as the fold increase in serum H5N1 HI antibody GMTs post-vaccination compared to Day 0, at Days 21 and 182. The H5N1 vaccine strain included A/Indonesia antigen.
Time Frame: At Day 21 and Day 182
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Increase
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Fold Increase
  A/Indonesia at Day 21 | 3.2 [2.2 to 4.6] | 2.8 [2.0 to 4.0]
  A/Indonesia at Day 182: number analyzed (Participants) | 49 | 50
  A/Indonesia at Day 182 | 5.1 [3.5 to 7.6] | 6.9 [5.1 to 9.2]

8. Secondary Outcome: Number of Subjects Seroprotected for H5N1 HI Antibodies
Description: A seroprotected subject was defined as a subject with a serum H5N1 HI antibody titer greater than or equal to 1:40, at Days 21 and 182. The H5N1 vaccine strain included A/Indonesia antigen.
Time Frame: At Day 0, Day 21 and Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  A/Indonesia at Day 0 | 0 | 0
  A/Indonesia at Day 21 | 19 | 16
  A/Indonesia at Day 182: number analyzed (Participants) | 49 | 50
  A/Indonesia at Day 182 | 29 | 38

9. Secondary Outcome: Antibody Titers for Serum Anti-H5N1 Neutralising Antibodies
Description: Antibody titers were expressed as Geometric mean titers (GMTs). The H5N1 vaccine strain included A/Indonesia antigen.
Time Frame: At Day 0, Day 42 and Day 182
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Titer
  A/Indonesia at Day 0: number analyzed (Participants) | 50 | 49
  A/Indonesia at Day 0 | 14.4 [13.6 to 15.2] | 18.3 [15.4 to 21.8]
  A/Indonesia at Day 42 | 579.6 [466.5 to 720.0] | 473.8 [379.9 to 591.0]
  A/Indonesia at Day 182: number analyzed (Participants) | 49 | 50
  A/Indonesia at Day 182 | 240.5 [210.3 to 275.0] | 240.1 [210.0 to 274.5]

10. Secondary Outcome: Number of Subjects Seroconverted for Serum Anti-H5N1 Neutralising Antibodies
Description: A seroconverted subject was defined as a subject with a minimum 4 fold increase in titer at post-vaccination for neutralising antibody response at Days 42 and 182.
  The H5N1 vaccine strain included A/Indonesia antigen.
Time Frame: At Day 42 and Day 182
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  A/Indonesia at Day 42: number analyzed (Participants) | 50 | 49
  A/Indonesia at Day 42 | 49 | 47
  A/Indonesia at Day 182: number analyzed (Participants) | 49 | 49
  A/Indonesia at Day 182 | 48 | 44

11. Secondary Outcome: Number of Subjects With Any Biochemical and Haematological Laboratory Abnormalities
Description: Biochemical and haematological parameters assessed in blood samples include alanine aminotransferase (ALT), aspartate aminotransferase (AST), basophils (BAS) and blood urea nitrogen (BUN ). Categories = unknown, below, within, or above the normal ranges.
Time Frame: At Day 0, Day 7 and Day 42
Population: Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  ALT [Unknown] at Day 0 | 0 | 0
  ALT [Unknown] at Day 7 | 0 | 0
  ALT [Unknown] at Day 42 | 0 | 0
  ALT [Below] at Day 0 | 0 | 0
  ALT [Below] at Day 7 | 1 | 0
  ALT [Below] at Day 42 | 1 | 0
  ALT [Within] at Day 0 | 47 | 46
  ALT [Within] at Day 7 | 47 | 45
  ALT [Within] at Day 42 | 45 | 46
  ALT [Above] at Day 0 | 3 | 4
  ALT [Above] at Day 7 | 2 | 5
  ALT [Above] at Day 42 | 4 | 4
  AST [Unknown] at Day 0 | 0 | 0
  AST [Unknown] at Day 7 | 0 | 0
  AST [Unknown] at Day 42 | 0 | 0
  AST [Below] at Day 0 | 0 | 0
  AST [Below] at Day 7 | 0 | 0
  AST [Below] at Day 42 | 0 | 0
  AST [Within] at Day 0 | 49 | 49
  AST [Within] at Day 7 | 50 | 49
  AST [Within] at Day 42 | 49 | 50
  AST [Above] at Day 0 | 1 | 1
  AST [Above] at Day 7 | 0 | 1
  AST [Above] at Day 42 | 1 | 0
  BAS [Unknown] at Day 0 | 0 | 0
  BAS [Unknown] at Day 7 | 0 | 0
  BAS [Unknown] at Day 42 | 0 | 0
  BAS [Below] at Day 0 | 0 | 0
  BAS [Below] at Day 7 | 0 | 0
  BAS [Below] at Day 42 | 0 | 0
  BAS [Within] at Day 0 | 50 | 49
  BAS [Within] at Day 7 | 50 | 50
  BAS [Within] at Day 42 | 50 | 50
  BAS [Above] at Day 0 | 0 | 1
  BAS [Above] at Day 7 | 0 | 0
  BAS [Above] at Day 42 | 0 | 0
  BUN [Unknown] at Day 0 | 0 | 0
  BUN [Unknown] at Day 7 | 0 | 0
  BUN [Unknown] at Day 42 | 0 | 0
  BUN [Below] at Day 0 | 0 | 1
  BUN [Below] at Day 7 | 0 | 0
  BUN [Below] at Day 42 | 1 | 0
  BUN [Within] at Day 0 | 50 | 48
  BUN [Within] at Day 7 | 50 | 50
  BUN [Within] at Day 42 | 49 | 49
  BUN [Above] at Day 0 | 0 | 1
  BUN [Above] at Day 7 | 0 | 0
  BUN [Above] at Day 42 | 0 | 1

12. Secondary Outcome: Number of Subjects With Any Biochemical and Haematological Laboratory Abnormalities
Description: Biochemical and haematological parameters assessed in blood samples include creatinine (CREA), eosinophils (EOS), hemoglobin (HB) and hematocrit (HC).
  Categories = unknown, below, within, or above the normal ranges.
Time Frame: At Day 0, Day 7 and Day 42
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  CREA [Unknown] at Day 0 | 0 | 0
  CREA [Unknown] at Day 7 | 0 | 0
  CREA [Unknown] at Day 42 | 0 | 0
  CREA [Below] at Day 0 | 1 | 2
  CREA [Below] at Day 7 | 1 | 3
  CREA [Below] at Day 42 | 2 | 3
  CREA [Within] at Day 0 | 48 | 44
  CREA [Within] at Day 7 | 46 | 44
  CREA [Within] at Day 42 | 47 | 45
  CREA [Above] at Day 0 | 1 | 4
  CREA [Above] at Day 7 | 3 | 3
  CREA [Above] at Day 42 | 1 | 2
  EOS [Unknown] at Day 0 | 0 | 0
  EOS [Unknown] at Day 7 | 0 | 0
  EOS [Unknown] at Day 42 | 0 | 0
  EOS [Below] at Day 0 | 0 | 0
  EOS [Below] at Day 7 | 0 | 0
  EOS [Below] at Day 42 | 0 | 0
  EOS [Within] at Day 0 | 44 | 46
  EOS [Within] at Day 7 | 45 | 46
  EOS [Within] at Day 42 | 47 | 46
  EOS [Above] at Day 0 | 6 | 4
  EOS [Above] at Day 7 | 5 | 4
  EOS [Above] at Day 42 | 3 | 4
  HB [Unknown] at Day 0 | 0 | 0
  HB [Unknown] at Day 7 | 0 | 0
  HB [Unknown] at Day 42 | 0 | 0
  HB [Below] at Day 0 | 1 | 4
  HB [Below] at Day 7 | 1 | 4
  HB [Below] at Day 42 | 2 | 5
  HB [Within] at Day 0 | 49 | 45
  HB [Within] at Day 7 | 49 | 44
  HB [Within] at Day 42 | 48 | 44
  HB [Above] at Day 0 | 0 | 1
  HB [Above] at Day 7 | 0 | 2
  HB[Above] at Day 42 | 0 | 1
  HC [Unknown] at Day 0 | 0 | 0
  HC [Unknown] at Day 7 | 0 | 0
  HC[Unknown] at Day 42 | 0 | 0
  HC [Below] at Day 0 | 0 | 1
  HC [Below] at Day 7 | 0 | 1
  HC [Below] at Day 42 | 0 | 1
  HC [Within] at Day 0 | 50 | 45
  HC [Within] at Day 7 | 50 | 46
  HC [Within] at Day 42 | 49 | 44
  HC [Above] at Day 0 | 0 | 4
  HC [Above] at Day 7 | 0 | 3
  HC [Above] at Day 42 | 1 | 5

13. Secondary Outcome: Number of Subjects With Any Biochemical and Haematological Laboratory Abnormalities
Description: Biochemical and haematological parameters assessed in blood samples include lymphocytes (LYM), monocytes (MON) and neutrophils (NEU).
  Categories = unknown, below, within, or above the normal ranges.
Time Frame: At Day 0, Day 7 and Day 42
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  LYM [Unknown] at Day 0 | 0 | 0
  LYM [Unknown] at Day 7 | 0 | 0
  LYM [Unknown] at Day 42 | 0 | 0
  LYM [Below] at Day 0 | 0 | 2
  LYM [Below] at Day 7 | 0 | 1
  LYM [Below] at Day 42 | 5 | 1
  LYM [Within] at Day 0 | 50 | 48
  LYM [Within] at Day 7 | 50 | 49
  LYM [Within] at Day 42 | 45 | 49
  LYM [Above] at Day 0 | 0 | 0
  LYM [Above] at Day 7 | 0 | 0
  LYM [Above] at Day 42 | 0 | 0
  MON [Unknown] at Day 0 | 0 | 0
  MON [Unknown] at Day 7 | 0 | 0
  MON [Unknown] at Day 42 | 0 | 0
  MON [Below] at Day 0 | 0 | 0
  MON [Below] at Day 7 | 0 | 0
  MON [Below] at Day 42 | 0 | 0
  MON [Within] at Day 0 | 50 | 49
  MON [Within] at Day 7 | 48 | 49
  MON [Within] at Day 42 | 49 | 50
  MON [Above] at Day 0 | 0 | 1
  MON [Above] at Day 7 | 2 | 1
  MON [Above] at Day 42 | 1 | 0
  NEU [Unknown] at Day 0 | 0 | 0
  NEU [Unknown] at Day 7 | 0 | 0
  NEU [Unknown] at Day 42 | 0 | 0
  NEU [Below] at Day 0 | 0 | 0
  NEU [Below] at Day 7 | 1 | 1
  NEU [Below] at Day 42 | 0 | 0
  NEU [Within] at Day 0 | 50 | 48
  NEU [Within] at Day 7 | 48 | 48
  NEU [Within] at Day 42 | 46 | 49
  NEU [Above] at Day 0 | 0 | 2
  NEU [Above] at Day 7 | 1 | 1
  NEU [Above] at Day 42 | 4 | 1

14. Secondary Outcome: Number of Subjects With Any Biochemical and Haematological Laboratory Abnormalities
Description: as for outcome 13
Time Frame: At Day 0, Day 7 and Day 42
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group. | Influenza A (H5N1) 41-64 Years Group.
Number analyzed (Participants) | 50 | 50
Participants
  PLA [Unknown] at Day 0 | 0 | 2
  PLA [Unknown] at Day 7 | 0 | 1
  PLA [Unknown] at Day 42 | 0 | 0
  PLA [Below] at Day 0 | 0 | 0
  PLA [Below] at Day 7 | 0 | 0
  PLA [Below] at Day 42 | 0 | 0
  PLA [Within] at Day 0 | 50 | 48
  PLA [Within] at Day 7 | 50 | 48
  PLA [Within] at Day 42 | 50 | 50
  PLA [Above] at Day 0 | 0 | 0
  PLA [Above] at Day 7 | 0 | 1
  PLA [Above] at Day 42 | 0 | 0
  RBC [Unknown] at Day 0 | 0 | 0
  RBC [Unknown] at Day 7 | 0 | 0
  RBC[Unknown] at Day 42 | 0 | 0
  RBC [Below] at Day 0 | 2 | 1
  RBC [Below] at Day 7 | 2 | 1
  RBC [Below] at Day 42 | 2 | 0
  RBC [Within] at Day 0 | 48 | 47
  RBC [Within] at Day 7 | 48 | 46
  RBC [Within] at Day 42 | 46 | 48
  RBC [Above] at Day 0 | 0 | 2
  RBC[Above] at Day 7 | 0 | 3
  RBC[Above] at Day 42 | 2 | 2
  WBC[Unknown] at Day 0 | 0 | 0
  WBC [Unknown] at Day 7 | 0 | 0
  WBC [Unknown] at Day 42 | 0 | 0
  WBC [Below] at Day 0 | 2 | 2
  WBC [Below] at Day 7 | 1 | 1
  WBC [Below] at Day 42 | 1 | 1
  WBC [Within] at Day 0 | 47 | 46
  WBC [Within] at Day 7 | 49 | 48
  WBC [Within] at Day 42 | 47 | 47
  WBC [Above] at Day 0 | 1 | 2
  WBC [Above] at Day 7 | 0 | 1
  WBC [Above] at Day 42 | 2 | 2

15. Secondary Outcome: Number of Subjects With Any Normal or Abnormal Urine Values
Description: Urine parameters assessed were blood, glucose, protein and urobilinogen. Categories = negative, positive
Time Frame: At Day 0, Day 7 and Day 42
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  Blood [Negative] at Day 0 | 48 | 44
  Blood [Positive] at Day 0 | 2 | 6
  Blood [Negative] at Day 7 | 47 | 43
  Blood [Positive] at Day 7 | 3 | 7
  Blood [Negative] at Day 42 | 46 | 46
  Blood [Positive] at Day 42 | 4 | 4
  Glucose [Negative] at Day 0 | 50 | 49
  Glucose [Positive] at Day 0 | 0 | 1
  Glucose [Negative] at Day 7 | 50 | 47
  Glucose [Positive] at Day 7 | 0 | 3
  Glucose [Negative] at Day 42 | 50 | 49
  Glucose [Positive] at Day 42 | 0 | 1
  Protein [Negative] at Day 0 | 49 | 50
  Protein [Positive] at Day 0 | 1 | 0
  Protein [Negative] at Day 7 | 48 | 50
  Protein [Positive] at Day 7 | 2 | 0
  Protein [Negative] at Day 42 | 49 | 49
  Protein [Positive] at Day 42 | 1 | 1
  Urobilinogen [Negative] at Day 0 | 47 | 50
  Urobilinogen [Positive] at Day 0 | 3 | 0
  Urobilinogen [Negative] at Day 7 | 49 | 50
  Urobilinogen [Positive] at Day 7 | 1 | 0
  Urobilinogen [Negative] at Day 42 | 49 | 50
  Urobilinogen [Positive] at Day 42 | 1 | 0

16. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling/induration. Any=any solicited local symptom reported regardless of their intensity. Grade 3 pain= significant pain at rest that prevented normal activities as assessed by inability to attend/do work or school. Grade 3 redness and swelling/induration=redness and swelling/induration above 100 millimetres (mm).
Time Frame: During the 7-day post vaccination period (Days 0-6) after any vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  Any Pain | 49 | 49
  Grade 3 Pain | 1 | 0
  Any redness | 12 | 16
  Grade 3 redness | 2 | 2
  Any swelling/induration | 17 | 23
  Grade 3 swelling/induration | 3 | 2

17. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were fatigue, headache, joint pain, muscle aches, shivering, increase sweating and fever. Any=any solicited general symptom reported regardless of their intensity grade or their relationship to vaccination. Any fever was ≥ 38.0 degrees celsius (°C). Grade 3 = general symptom that prevented normal everyday activities as assessed by inability to attend/do work or school, or required intervention of a physician/healthcare provider. Grade 3 fever was≥ 39.0°C. Related= general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day post vaccination period (Days 0-6) after any vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  Any fatigue | 39 | 32
  Grade 3 fatigue | 3 | 0
  Related fatigue | 39 | 32
  Any headache | 30 | 21
  Grade 3 headache | 0 | 0
  Related headache | 27 | 21
  Any joint pain | 16 | 18
  Grade 3 joint pain | 1 | 0
  Related joint pain | 16 | 17
  Any muscle aches | 36 | 34
  Grade 3 muscle aches | 1 | 0
  Related muscle aches | 36 | 33
  Any shivering | 13 | 7
  Grade 3 shivering | 2 | 0
  Related shivering | 11 | 7
  Any increase sweating | 13 | 8
  Grade 3 increase sweating | 0 | 0
  Related increase sweating | 12 | 8
  Any fever | 6 | 5
  Grade 3 fever | 1 | 0
  Related fever | 6 | 5

18. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE is any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the 21-day (Days 0-20) following vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  Any unsolicited AE (s) | 27 | 24
  Grade 3 unsolicited AE (s) | 3 | 0
  Related unsolicited AE (s) | 11 | 17

19. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs
Description: as for outcome 18
Time Frame: From Day 0 to Day 83 following vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants
  Any unsolicited AE (s) | 33 | 36
  Grade 3 unsolicited AE (s | 3 | 2
  Related unsolicited AE (s) | 11 | 17

20. Secondary Outcome: Number of Subjects Reporting Any Medically-significant Conditions (MSCs)
Description: MSCs were defined as AEs with a medically-attended visit (s) i.e. prompting emergency room (ER) visits, hospitalizations or physician visits and that were not routine visits for physical examination or vaccination.
Time Frame: During the 182-day (Days 0-181) post-vaccination period
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants | 34 | 26

21. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (Day 0 to Day 181)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Number analyzed (Participants) | 50 | 50
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events = From Days 0-181. Systematically assessed frequent adverse events (AEs) = During the 7 day post vaccination period. Non-systematically assessed frequent AEs= During Days 0-20 and Days 0-84 post vaccination period respectively.
Arm/Group | Influenza A (H5N1) 20-40 Years Group | Influenza A (H5N1) 41-64 Years Group
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 50/50 | 50/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza A (H5N1) 20-40 Years Group (N=50) | Influenza A (H5N1) 41-64 Years Group (N=50)
Pain (General disorders) | 49 | 49
Redness (General disorders) | 12 | 16
Swelling/ Induration (General disorders) | 17 | 23
Fatigue (General disorders) | 39 | 32
Headache (General disorders) | 30 | 21
Joint pain (General disorders) | 16 | 18
Muscle aches (General disorders) | 36 | 34
Shivering (General disorders) | 13 | 7
Increase Sweating (General disorders) | 13 | 8
Fever (General disorders) | 6 | 5
Injection site pruritus (General disorders) | 5 | 9 — Assessed during Days 0-20 post vaccination period
Injection site warmth (General disorders) | 6 | 8 — Assessed during Days 0-20 post vaccination period
Nasopharyngitis (Infections and infestations) | 7 | 1 — Assessed during Days 0-20 post vaccination period
Diarrhoea (Gastrointestinal disorders) | 3 | 0 — Assessed during Days 0-20 post vaccination period
Injection site pruritus (General disorders) | 5 | 9 — Assessed during Days 0-83 post vaccination period
Nasopharyngitis (Infections and infestations) | 9 | 8 — Assessed during Days 0-83 post vaccination period
Injection site warmth (General disorders) | 6 | 8 — Assessed during Days 0-83 post vaccination period
Headache (Nervous system disorders) | 3 | 6 — Assessed during Days 0-83 post vaccination period
Bronchitis (Infections and infestations) | 5 | 1 — Assessed during Days 0-83 post vaccination period
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 — Assessed during Days 0-83 post vaccination period
Diarrhoea (Gastrointestinal disorders) | 3 | 0 — Assessed during Days 0-83 post vaccination period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.